CLINICAL TRIAL: NCT01416077
Title: Perioperative Goal Directed Fluid Therapy During Esophageal Resection A Prospective Randomized Controlled Open Multi-centre Trial to Study the Effect on Postoperative Complications
Brief Title: Decreasing Postoperative Complications by Goal-Directed Fluid Therapy During Esophageal Resection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Lena Nilsson, MD pHd, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USANOP001
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Esophageal Cancer
Keywords: fluid; goal-directed; FloTrac; pulse contour analysis; postoperative complications; anesthesia; esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard treatment (No Intervention): Fluid and inotropic drugs are given based on conventional parameters such as blood pressure and heart rate as judged by the individual anesthesiologists judgement.
- goal-directed fluid treatment (Active Comparator): Stroke Volume and Cardiac Index are measured with the Flotrac/Vigileo system and circulation is optimised
  Interventions: Other: fluid optimisation

INTERVENTIONS:
Other: fluid optimisation — Stroke Volume and Cardiac Index are measured with the Flotrac/Vigileo system and circulation is optimised
  1. Crystalloid infusion (2,5 ml/kg/t) throughout surgery
  2. 3 ml/kg Volulyte (synthetic colloid) is infused during 5 minutes and SV is measured directly before and 5 minutes after. If SV increases more than 10% the dose is repeated until no increase > 10% is observed. A new dose is given if SV decreases more than 10% from the last value.
  3. If despite optimal filling Cardiac Index (CI) is below 2,5 l/min/m2 infusion with dobutamin is started to attain CI > 2,5.
  4. If despite CI > 2,5 Mean Arterial Pressure <65 mmHg vasopressor (phenylephrine / norepinephrine) is started until MAP equals or is over 65.
  Arms: goal-directed fluid treatment

SUMMARY:
Surgery for cancer of the esophagus is associated with a high risk of postoperative complications. It has been shown that the risk of postoperative complications can be decreased by optimising the amount and type of infusion fluids given during surgery, steered by measurement of cardiac stroke volume, mostly done with a device called esophageal Doppler. This device can however not be used during this type of surgery. This study wants to test the hypothesis that postoperative complications in patients operated for esophageal cancer can be partially prevented by using a goal directed strategy for the administration of fluids and drugs influencing the heart and vessels, based on measurement of stroke volume by pulse wave analysis (FloTrac).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for transthoracic esophageal resection because of malignancy, without colonic interposition who leave informed consent

Exclusion Criteria:

* ASA 4 or 5
* Atrial Fibrillation
* Significant Aortic or Mitral Valve Insufficiency
* Preoperative planned extensive monitoring beyond CVP, arterial blood pressure, diuresis, ECG and other standard monitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Incidence of complications 5 and 30 days postoperatively | 5 and 30 days postoperatively

SECONDARY OUTCOMES:
length of stay ICU and total hospital | 30 days
return of bowel function | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Lena Nilsson, MD PhD, Study Chair — University Hospital, Linkoeping
Locations (1):
- University Hospital Linkoeping, Linköping, Sweden

REFERENCES:
- [Background] Bahlmann H, Halldestam I, Nilsson L. Goal-directed therapy during transthoracic oesophageal resection does not improve outcome: Randomised controlled trial. Eur J Anaesthesiol. 2019 Feb;36(2):153-161. doi: 10.1097/EJA.0000000000000908. PMID 30431499